CLINICAL TRIAL: NCT05563311
Title: Functional Assessment and Sleep Apnea in Obese Children and Adolescents After a Telerehabilitation Program
Brief Title: Functional Assessment and Sleep Apnea in Obese Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, LUCIANA MARIA MALOSA SAMPAIO, Clinical Professor, University of Nove de Julho
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Obese Children and Adolescents
Record Dates: First submitted 2022-09-26; First posted 2022-10-03 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Obstructive Sleep Apnea; Balance; Obesity, Childhood
Keywords: pediatric obesity; pediatric obstructive sleep apnea; Postural balance
MeSH Terms: conditions — Sleep Apnea, Obstructive; Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- high-intensity interval training (Experimental): High-intensity interval training describes physical exercise that is characterized by brief, intermittent bursts of vigorous activity, interspersed with periods of rest or low-intensity exercise
  Interventions: Other: Exercise on High-intensity interval training

INTERVENTIONS:
Other: Exercise on High-intensity interval training — 3 times a week, for 8 weeks

SUMMARY:
Childhood obesity increases significantly, and determines several complications in childhood and adulthood, and the worldwide prevalence of childhood obesity has shown a rapid increase in recent decades.

The severity of obesity-related risk factors is directly linked to body fat topography, and variations in body fat distribution in obese children can be of high value in predicting future health risks, like of cardiovascular disease in adulthood.

There is a potential correlation between obesity and sleep disorders, increasing the predisposition to obstructive sleep apnea syndrome, that is a frequent complication, affecting up to 80% of obese children and adolescents.

In relation to postural control, and that anthropometric indicators interfere with children's postural balance, already verified by balance assessment using computerized dynamic posturography.

Several studies show that physical activity in childhood and adolescence can influence healthy habits in adulthood. Children and youth ages 5 to 17 should accumulate at least 60 minutes of moderate to vigorous-intensity physical activity daily.

It is important to emphasize that the COVID-19 has impacted every aspect of healthcare delivery, and therefore Telerehabilitation has been satisfactorily addressed in reabilitation In the exercise recommendations for children, exercise programs performing aerobic and resistance exercises at a high level of intensity, on a frequent basis (3-5 days a week) for 30-80 minutes, seeking intensity of 50-90% of the maximum heart rate (HRmax), can be used and are shown to be efficient for the treatment of obesity. Therefore the High-intensity interval training (HIIT) describes physical exercise that is characterized by brief, intermittent bursts of vigorous activity, interspersed with periods of rest, cab generate favorable metabolic adaptations on sleep and body weight loss.

Outcome Measures:

Primary Outcome Measures

* The effects of high-intensity interval training (HIIT) and high-intensity functional training (HIFT) through Telerehabilitation on body composition and Obstructive sleep apnea (assessed by body mass index and bioimpedanceand polysomnography type 4) Secondary Outcome Measures
* Functional performance of children and adolescents (3 minute step test)
* Balance (balance assessments with Wii Balance board)

Inclusion Criteria:

* Age ≥ 6 to 17 years;
* Confirmed obesity children by body mass index acorrding to the age

DETAILED DESCRIPTION:
Outcome Measures:

Primary Outcome Measures

- The effects of high-intensity interval training (HIIT) and high-intensity functional training (HIFT) through Telerehabilitation on body composition and Obstructive sleep apnea (assessed by body mass index and bioimpedance and polysomnography type 4)

Secondary Outcome Measures

* Functional performance of children and adolescents (3 minute step test)
* Balance (balance assessments with Wii Balance board)

Inclusion Criteria:

* Age ≥ 6 to 17 years;
* Confirmed obesity children by body mass index acorrding to the age

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 6 to 17 years;

* Confirmed obesity children by body mass index acorrding to the age

Exclusion Criteria:

* orthopedic or neurological conditions that make it impossible to in a physical participation program

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Apnea hypopnea index | 1 day
  AHI

SECONDARY OUTCOMES:
Functional performance of children and adolescents (3 minute step test) | 1 day
  numbers steps
Balance (balance assessments with Wii Balance board) | 1 day
  COP

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Malosa, Study Director — University of Nove de Julho
Locations (1):
- Luciana Malosa, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Magalhaes EI, Sant'Ana LF, Priore SE, Franceschini Sdo C. [Waist circumference, waist/height ratio, and neck circumference as parameters of central obesity assessment in children]. Rev Paul Pediatr. 2014 Sep;32(3):273-81. doi: 10.1590/0103-0582201432320. Epub 2014 Oct 3. PMID 25479861
- [Background] Atar M, Pirgon O, Buyukgebiz A. Sleep Disorders and Obesity in Childhood: A New Component in Solving Obesity. Pediatr Endocrinol Rev. 2019 Jun;16(4):441-451. doi: 10.17458/per.vol16.2019.apb.sleepdisordersobesitychildhood. PMID 31245939
- [Background] Ye XH, Chen H, Kang XG, Zhang Q. [Association between obesity and sleep disorders among children in Lanzhou, China]. Zhongguo Dang Dai Er Ke Za Zhi. 2019 Oct;21(10):987-991. doi: 10.7499/j.issn.1008-8830.2019.10.007. Chinese. PMID 31642432
- [Background] Greve J, Alonso A, Bordini AC, Camanho GL. Correlation between body mass index and postural balance. Clinics (Sao Paulo). 2007 Dec;62(6):717-20. doi: 10.1590/s1807-59322007000600010. PMID 18209913
- [Background] Deforche BI, Hills AP, Worringham CJ, Davies PS, Murphy AJ, Bouckaert JJ, De Bourdeaudhuij IM. Balance and postural skills in normal-weight and overweight prepubertal boys. Int J Pediatr Obes. 2009;4(3):175-82. doi: 10.1080/17477160802468470. PMID 18972242
- [Background] Villarrasa-Sapina I, Alvarez-Pitti J, Cabeza-Ruiz R, Redon P, Lurbe E, Garcia-Masso X. Relationship between body composition and postural control in prepubertal overweight/obese children: A cross-sectional study. Clin Biomech (Bristol). 2018 Feb;52:1-6. doi: 10.1016/j.clinbiomech.2017.12.010. Epub 2017 Dec 21. PMID 29291461
- [Background] Feito Y, Heinrich KM, Butcher SJ, Poston WSC. High-Intensity Functional Training (HIFT): Definition and Research Implications for Improved Fitness. Sports (Basel). 2018 Aug 7;6(3):76. doi: 10.3390/sports6030076. PMID 30087252